CLINICAL TRIAL: NCT04353687
Title: PROGRESS: A PROspective Evaluation of the Early surGeon expeRiencE With Robotic-aSSisted (RA) Inguinal Hernia Repair (IHR)
Brief Title: Early Surgeon Experience With Robotic-Assisted Inguinal Hernia Repair
Status: Active, not recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-HLC-2019
Record Dates: First submitted 2020-04-09; First posted 2020-04-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Cohort 1 Open Surgeons: Primarily open inguinal hernia surgeon with no or limited previous robotic-assisted experience.
  Interventions: Device: Robotic-assisted inguinal hernia repair
- Cohort 2 Laparoscopic Surgeons: Primarily laparoscopic inguinal hernia surgeon with no or limited previous robotic-assisted experience.
  Interventions: Device: Robotic-assisted inguinal hernia repair

INTERVENTIONS:
Device: Robotic-assisted inguinal hernia repair — Each surgeon will perform the robotic-assisted inguinal hernia procedure per their standard practice. Surgeon subjects will consent to prospectively provide selected procedure and case data.

SUMMARY:
The primary objective of this study is to evaluate the progression of surgeon efficiency and proficiency of traditionally open or laparoscopic surgeons performing robotic-assisted inguinal hernia repair throughout their learning curve.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational pilot study evaluating surgeon efficiency and proficiency of traditionally open or laparoscopic surgeons performing robotic-assisted inguinal hernia repair. The study will focus on surgeon intraoperative efficiency and technical performance outcomes as well as conversions, intraoperative complications, and mental and cognitive workload. Surgeon subjects will be assessed for technical proficiency through a study specific technical proficiency form and the GEARS scale by independent surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent by adult surgeon subject
2. Practicing general surgeon with no or limited robotic assisted experience
3. Full access to the da Vinci surgical system at hospital and ability to perform robotic cases as needed
4. Willingness to participate in all aspects of the study

Exclusion Criteria:

1. Condition(s) that, in the opinion of the investigator, may prevent completion of the study or protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended study population will be compromised of general surgeons. All surgeons will be qualified general surgeons by training and experienced in performing open or laparoscopic inguinal hernia repair and will be transitioning to robotic-assisted inguinal hernia repair. All surgeons will have zero or minimal experience with robotic-assisted inguinal hernia repair.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of surgeon efficiency | Assessed intraoperatively (all cases)
  Change of skin to skin procedure time, dissection time, time to establish critical view of the myopectineal orifice (MPO), and mesh fixation time through the assessment of intraoperative tasks
Change of surgeon proficiency/performance | Within one month following surgery (every 12th case ± 2 cases)
  Change of technical proficiency scores and Global Evaluative Assessment of Robotic Skills (GEARS) scores cases as assessed by independent video review.

OTHER OUTCOMES:
Change in cognitive and mental workload (SURG-TLX) | With one hour following surgery (every 5th case ± 1 case)
  Change in cognitive and mental workload as assessed by the Surgery Task Load Index (SURG-TLX)
Change of surgeon efficiency | Assessed intraoperatively (all cases)
  Change of console time, docking time, and operative room time through the assessment of intraoperative tasks
Conversion to Open | Intraoperative
  Incidence of conversions of the robotic-assisted procedure
Number of Complications | Intraoperative and 30 days following discharge from hospital
  Intraoperative and post-operative complications related to the inguinal hernia repair
Length of hospital stay (LOS) | Arrival of the patient in the operating room to the time of patient discharge, up to an approximate of one week
  The length of patient admission to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside Hospital, Newport News, Virginia, United States

IPD SHARING:
Plan to Share IPD: No